CLINICAL TRIAL: NCT04126265
Title: Artificial Intelligence-assisted Colonoscopy for Detection of Colon Polyps: a Prospective Randomized Cohort Study
Brief Title: Artificial Intelligence-assisted Colonoscopy for Detection of Colon Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Side Liu (Other)
Responsible Party: Sponsor-Investigator, Side Liu, professor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NCT201908-K5-01
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Artificial Intelligence; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine colonoscopy group (No Intervention): The patient underwent routine colonoscopy.
- Artificial intelligence assisted colonoscopy group (Experimental): The real-time automatic polyp detection system was used to assist the endoscopist.
  Interventions: Device: Artificial intelligence assisted colonoscopy

INTERVENTIONS:
Device: Artificial intelligence assisted colonoscopy — The colonoscopy is connected to the real-time polyp detection system. If the polyp is detected by enteroscopy, the alarm will be given.
  Arms: Artificial intelligence assisted colonoscopy group

SUMMARY:
All subjects shall sign informed consent before screening, and subjects shall be included according to inclusion and exclusion criteria.

A total of four endoscopists were included in the study, two in each group of senior endoscopists and two in each group of junior endoscopists.

Patients were randomly enrolled into the senior endoscopy group and the junior endoscopy group, and received artificial intelligence assisted colonoscopy and conventional colonoscopy successively. The two colonoscopy methods were performed back to back by different endoscopy physicians with the same seniority.

All patients were examined and treated according to routine medical procedures. The routine colonoscopy group and the artificial-intelligence-assisted colonoscopy group made detailed records of the patients' withdrawal time, entry time, number of polyps detected, polyp Paris classification, polyp size, polyp shape, polyp location and intestinal preparation during the colonoscopy process

DETAILED DESCRIPTION:
This is a prospective randomized clinical study.This study was conducted in the Endoscopy Center of the Nanfang Hospital, China. Routine bowel preparation consisted of 4 L of polyethylene glycol, given in split doses. Colonoscopies were performed with high definition colonoscopes and high-definition monitors.

All subjects shall sign informed consent before screening, and subjects shall be included according to inclusion and exclusion criteria.

A total of four endoscopists were included in the study, two in each group of senior endoscopists (>1000 colonoscopies) and two in each group of junior endoscopists ( <1000 colonoscopies).

Patients were randomly enrolled into the senior endoscopy group and the junior endoscopy group, and received artificial intelligence assisted colonoscopy and conventional colonoscopy successively. The two colonoscopy methods were performed by different endoscopy physicians back to back with the same seniority.

All patients were examined and treated according to routine medical procedures (outpatient patients and inpatients who did not sign the consent form for polypectomy were not resected for the lesions detected during the examination, while inpatients who signed the consent form for polypectomy were left in the original position after the first colonoscopy and removed at the end of the second examination).

The routine colonoscopy group and the artificial-intelligence-assisted colonoscopy group made detailed records of the patients' withdrawal time, entry time, number of polyps detected, polyp Paris classification, polyp size, polyp shape, polyp location and intestinal preparation during the colonoscopy process.

ELIGIBILITY:
Inclusion Criteria:

Chinese population aged 18-80 years old; Patients voluntarily signed informed consent form; In accordance with the indications of colonoscopy.

Exclusion Criteria:

(IBD) history of inflammatory bowel disease; History of colorectal surgery; Previous failed colonoscopy; Polyposis syndrome; Highly suspected colorectal cancer (CRC)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of small polyps (diameter < 6mm) | 6 months
  In each group, the number of patients with small polyps was detected as a percentage of the total number of patients.

SECONDARY OUTCOMES:
Number of polyps detected | 6 months
  Number of polyps found in each group.
Polyp size | 6 months
  Average size of all polyps detected in each group.
Polyp morphology | 6 months
  Morphological classification of all polyps detected in each group.

CONTACTS AND LOCATIONS:
Overall Officials: side liu, doctor degree, Principal Investigator — Chief physician
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo Y, Zhang Y, Liu M, Lai Y, Liu P, Wang Z, Xing T, Huang Y, Li Y, Li A, Wang Y, Luo X, Liu S, Han Z. Artificial Intelligence-Assisted Colonoscopy for Detection of Colon Polyps: a Prospective, Randomized Cohort Study. J Gastrointest Surg. 2021 Aug;25(8):2011-2018. doi: 10.1007/s11605-020-04802-4. Epub 2020 Sep 23. PMID 32968933